CLINICAL TRIAL: NCT02887105
Title: Memory and Emotion in Acute and Chronic Phases of Cerebrovascular Accident
Acronym: MEMOIRE ET EMO
Status: Completed | Type: Observational
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Sponsor
Other Study IDs: PSS2012/MEMOIRE-DUCROCQ/MS
Record Dates: First submitted 2016-08-24; First posted 2016-09-01 (Estimated); Last update posted 2016-09-08 (Estimated); Status verified 2016-08

CONDITIONS: Cerebrovascular Accident
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients with cerebrovascular accident
  Interventions: Other: Standard neuropsychological assessment; Other: Brain MRI

INTERVENTIONS:
Other: Standard neuropsychological assessment
Other: Brain MRI

SUMMARY:
The purpose is to determine the relationship between anxiety and cognitive performances in patients with acute and chronic phases of cerebrovascular accident (CVA). Data from neuropsychological assessment concerning cognitive processes (working and episodic memory) sensitive to different dimensions of anxiety will be analyzed.

The secondary purpose is to evaluate how some neurological (hemispherical lateralization of lesions), psychological (depression) and demographic (quality of life) variables can increase the effects of different dimensions of anxiety on cognitive processes, during the acute and/or chronic phase of CVA.

DETAILED DESCRIPTION:
Data will be collected during usual neuropsychological evaluation and cerebral imagery examination (NIHSS, Rankin scale) of patients in acute (0-1 month) and chronic (6 months) phases of CVA.

ELIGIBILITY:
Inclusion Criteria:

* Acute phase of carotid, vertebrobasilar or lacunar cerebrovascular accident with ischemic or hemorrhagic origin
* Right-handed
* Possible cooperation: understanding of French instructions
* Normal or corrected vision
* Normal or corrected hearing
* Mini-mental state examination score higher than pathologic threshold according to age and sociocultural level of patient
* Possible follow up of patient

Exclusion Criteria:

* Hearing problems
* Vision problems
* Right hemiplegia or acute monoparesis of right upper limb
* Hemispatial neglect
* Apraxia
* Psychiatric or neurological history possibly interfering with neuropsychological evaluation
* Important defect of working memory or executive functions

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients hospitalized for a cerebrovascular accident
Sampling Method: Non-Probability Sample
Enrollment: 76 (Actual)
Dates: Start 2012-12; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
State of anxiety evaluated with STAI-YA scale | up to 1 month (from CVA)
State of anxiety evaluated with STAI-YA scale | 6 months (from CVA)
Anxiety proneness evaluated with STAI-YB scale | up to 1 month (from CVA)
Anxiety proneness evaluated with STAI-YB scale | 6 months (from CVA)
Apprehension anxiety evaluated with Penn State Worry Questionnaire | up to 1 month (from CVA)
Apprehension anxiety evaluated with Penn State Worry Questionnaire | 6 months (from CVA)
Evaluation of working memory updating with N-back verbal and visuospatial task | up to 1 month (from CVA)
Evaluation of working memory updating with N-back verbal and visuospatial task | 6 months (from CVA)
Evaluation of working memory inhibition with Stimulus-response compatibility task | up to 1 month (from CVA)
Evaluation of working memory inhibition with Stimulus-response compatibility task | 6 months (from CVA)
Evaluation of working memory flexibility with Switching task | up to 1 month (from CVA)
Evaluation of working memory flexibility with Switching task | 6 months (from CVA)
Evaluation of verbal working memory with Wechsler memory scale | up to 1 month (from CVA)
Evaluation of verbal working memory with Wechsler memory scale | 6 months (from CVA)
Evaluation of visuospatial working memory with Wechsler memory scale | up to 1 month (from CVA)
Evaluation of visuospatial working memory with Wechsler memory scale | 6 months (from CVA)
Evaluation of visual episodic memory with Rey and Taylor figure test | 6 months (from CVA)
Evaluation of verbal episodic memory with RL/RI 16 item test | 6 months (from CVA)

SECONDARY OUTCOMES:
Hemispheric lateralization of lesions detected with MRI | up to 1 month from CVA
Depression state evaluated with Back depression inventory | up to 1 month (from CVA)
Depression state evaluated with Back depression inventory | 6 months (from CVA)
Quality of life evaluated with SF-36 test | after 6 months from CVA

CONTACTS AND LOCATIONS:
Overall Officials: Xavier DUCROCQ, Pr, Principal Investigator — Service de Neurologie - Unité Neurovasculaire - Hôpital Central Nancy
Locations (2):
- France (2):
  - Service de Neurologie - Hôpital Bon Secours - CHR de Metz-Thionville, Metz
  - Service de Neurologie - Hôpital Central - CHU de Nancy, Nancy